CLINICAL TRIAL: NCT03163069
Title: Does Use of a Whitening Dentifrice Improve the Efficiency of In-office Tooth Bleaching Procedures? A Double-blind Randomized Controlled Clinical Trial.
Brief Title: The Effect of Whitening Toothpaste on Tooth Color Associated With Bleaching Process
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Hao Yu, Fujian Medical University, Fujian Medical University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 20170318
Record Dates: First submitted 2017-05-16; First posted 2017-05-22 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Tooth Discoloration
Keywords: tooth bleaching; dentifrice
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Intervention Model Description: factorial assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Whitening dentifrice (Experimental): in-office bleaching with the conventional whitening dentifrice
  Interventions: Combination Product: in-office bleaching with the conventional whitening dentifrice
- Whitening dentifrice containing blue covarine (Experimental): in-office bleaching with the whitening dentifrice containing blue covarine
  Interventions: Combination Product: in-office bleaching with the whitening dentifrice containing blue covarine
- Regular dentifrice (Experimental): in-office bleaching with the regular dentifrice
  Interventions: Combination Product: in-office bleaching with the regular dentifrice

INTERVENTIONS:
Combination Product: in-office bleaching with the conventional whitening dentifrice — Participants will receive in-office tooth bleaching with 40% hydrogen peroxide (Opalescence Boost PF 40%) for the maxillary anterior teeth (2 sessions, with a 1-week interval). During the tooth bleaching procedure and 3 weeks after the procedure, the participants will be instructed to brush their teeth twice with the conventional whitening dentifrice.
  Arms: Conventional Whitening dentifrice
Combination Product: in-office bleaching with the whitening dentifrice containing blue covarine — Participants will receive in-office tooth bleaching with 40% hydrogen peroxide (Opalescence Boost PF 40%) for the maxillary anterior teeth (2 sessions, with a 1-week interval). During the tooth bleaching procedure and 3 weeks after the procedure, the participants will be instructed to brush their teeth twice with the whitening dentifrice containing blue covarine.
  Arms: Whitening dentifrice containing blue covarine
Combination Product: in-office bleaching with the regular dentifrice — Participants will receive in-office tooth bleaching with 40% hydrogen peroxide (Opalescence Boost PF 40%) for the maxillary anterior teeth (2 sessions, with a 1-week interval). During the tooth bleaching procedure and 3 weeks after the procedure, the participants will be instructed to brush their teeth twice with the regular dentifrice.
  Arms: Regular dentifrice

SUMMARY:
This double-blind randomized controlled clinical trial aimed to investigate the effect of whitening dentifrices on the clinical efficiency of in-office tooth bleaching procedures.

DETAILED DESCRIPTION:
Sixty-three eligible participants (29 males and 34 females, mean age 26.1 years) with at least one maxillary tooth demonstrating shade A3 or darker will be recruited and randomly allocated into 3 groups (n = 21), according to the different dentifrices used in this clinical trial: Crest Total (regular dentifrice) for group C, Crest 3D Whitening (conventional whitening dentifrice) for group CW, and Close Up White Now (whitening dentifrice containing blue covarine) for group CU. All participants will receive in-office tooth bleaching with 40% hydrogen peroxide (Opalescence Boost PF 40%) for the maxillary anterior teeth (2 sessions, with a 1-week interval). The participants will be instructed to use only the provided dentifrices and toothbrushes to brush their teeth twice daily over a 4-week period. Colour parameters (CIE L*, a*, b*) will be measured with a spectrophotometer (Vita Easyshade Advance 4.0) at baseline (T1), after the first bleaching session (T2), after the second bleaching session (T3), 1 week after the completion of in-office bleaching (T4), and 3 weeks after the completion of in-office bleaching (T5). The colour differences (ΔE) and whiteness index (W) will also be calculated. The data will be statistically analysed through repeated ANOVA and Tukey's test (α = 0.05).

ELIGIBILITY:
Inclusion Criteria:

* patients between 18 and 60 years of age, with fully erupted upper and lower incisors and canines without dental or periodontal disease or restorations, and with at least one maxillary tooth presenting color score A3 or darker, as measured with the Vita Classical guide (Vita Zahnfabrik, Bad Sa ̈ ckingen, Germany) ordered by brightness

Exclusion Criteria:

* patients with systemic diseases or oral mucosal disorders, previous bleaching treatment, patients undergoing orthodontic treatment, pregnant women, people with known allergy to the product ingredients, smokers, and alcohol abusers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2017-07-02 (Actual); Study Completion 2017-08-24 (Actual)

PRIMARY OUTCOMES:
Change in tooth colour | 4 weeks
  Colour parameters (CIE L*, a*, b*) will be measured with a spectrophotometer (Vita Easyshade Advance 4.0). The color alteration after each session will be given by the differences between the values obtained at the sessions and the baseline (∆E).

SECONDARY OUTCOMES:
Change in tooth whiteness | 4 weeks
  The whiteness index will be registered at the sessions and the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Yu, Principal Investigator — Fujian Medical University, China
Locations (1):
- Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided